CLINICAL TRIAL: NCT04207892
Title: PedORTHO-A Prospective Multicenter Observational Registry of Pediatric Orthopedic Trauma and Health Outcomes in Skeletally Immature Children
Brief Title: Registry of Pediatric Orthopedic Trauma and Health Outcomes in Skeletally Immature Children
Status: Active, not recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: PedORTHO
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Long Bone Fractures
MeSH Terms: interventions — Therapeutics; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Conservative (non-surgical) treatment — Cast Sling Splint Collar
Procedure: Surgical treatment — Elastic Stable Intramedullary Nailing (ESIN) K-Wire External fixation

SUMMARY:
International registry to collect prospective treatment and outcomes data on specific, key non-pathological fractures in children with open physes. Data will be collected during follow-up visits according to standard of care at 3 to 8 weeks, 3, 6, 12 and 24 months

DETAILED DESCRIPTION:
This international registry will collect prospective treatment and outcomes data on specific, key non-pathological fractures in children with open physes. The long-term goal is to build this registry to include all fractures according to the AO pediatric fracture classification (AO PCCF). However, to establish proof-of-principle and study feasibility, the investigators aim to first begin with the inclusion of a limited number of key long bone fracture types for which optimal treatment and management are under particular debate, or for which substantial clinical equipoise exists. Consequently, the investigators aim to begin with separate registry arms based on defined fracture segments in specific bones. Each registry arm will be defined by a customized set of outcomes to be collected. Participants will be enrolled into these specific arms according to their injury diagnosis. The registry arms will be categorized as follows:

* Proximal humerus fractures
* Distal humerus fractures
* Proximal radius fractures
* Forearm shaft fractures
* Tibial shaft fractures (with/without fibula fracture)

All participants enrolled in the registry will be followed over the course of their treatment from the time of enrolment to end of treatment in accordance with the treating surgeon's regular clinical practice. All relevant information will be recorded at baseline and at each follow-up visit that participants attend at the orthopedic clinic, according to standard of care for each fracture type. A standardized set of prospective data including demographic information, baseline injury information, diagnosis, treatment details and clinical, radiographic, functional, and PROs will be collected for each participant. Data involving additional outcomes or variables may also be collected depending on the specific sub-study or registry arm that the participant is enrolled in.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed open physis in the injured bone at time of injury
* Diagnosis of an isolated fracture according to the AO PCCF
* Willingness and ability of the patient/parents/legally responsible care giver to participate in the registry, including obtaining imaging and adhering to follow-up procedures according to standard of care in each clinic
* Willingness and ability of the parent(s) to support the patient in his/her study participation
* Ability of parents or a legal guardian to understand the content of the patient information/ICF and to sign and date the IRB/EC approved written informed consent form

Exclusion Criteria:

* Radiologically confirmed closed physis in the injured bone at time of injury
* Polytrauma/multiple fractures
* Previous fracture of the same anatomical region
* Underlying musculoskeletal or neuromuscular disorder
* Present to participating centers with a displaced humeral fracture, tibial shaft fracture, forearm fracture, or femoral neck fracture at greater than 4 weeks postinjury
* Unable to provide the legal consent
* Inability of the patient/parents/legally responsible caregiver to participate in imaging and/or FU procedures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Consecutive pediatric patients with key long bone fractures.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection of fracture and trauma details | up to 24 months
  To analyze the AO Pediatric Long Bone Fracture Classification in terms of utility for treatment decision-making and prediction of fracture outcomes

SECONDARY OUTCOMES:
Axial deviation and range of motion (ROM) | up to 24 months
  Axial deviation or difference in ROM in the shoulder (abduction/adduction, internal rotation/external rotation, flexion/extension), elbow (flexion/extension, varus/valgus), wrist (flexion/extension, abduction/adduction, supination/pronation), hip (flexion/extension, abduction/adduction, internal rotation/external rotation (in flexion)), knee (flexion/extension), ankle (flexion/extension, supination/pronation, abduction/adduction)
Leg length discrepancy | up to 24 months
  The Leg Length Discrepancy (LLD) will be measured using the standing blocks method
Return to full activity | up to 24 months
  Time to full weight-bearing, time to full activity, and time to return to kindergarten/school
Implant removal | up to 24 months
  Assessment if implant removal was done.
Patient-reported outcome | up to 24 months
  Patient Reported Outcomes of Fracture Healing

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, Prof, Principal Investigator — BC Children's Hospital, Vancouver; Emily Schaeffer, Dr, Principal Investigator — BC Children's Hospital, Vancouver; Alexander Joeris, Prof, Principal Investigator — AO foundation
Locations (17):
- University of Missouri Health Care, Columbia, Missouri, United States
- Australia (2):
  - Queensland Children's Hospital, Brisbane, Queensland
  - The Children's Hospital at Westmead, Sydney
- Canada (4):
  - IWK Health Centre, Halifax
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa
  - The Hospital for Sick Children, Toronto
  - BC Children's Hospital, Vancouver
- Hospital Base Valdivia, Valdivia, Chile
- Clinical Hospital Centre Rijeka, Rijeka, Croatia
- Kinderchirurgische Klinik, Klinikum Karlsruhe, Karlsruhe, Germany
- Tamale Teaching Hospital, Tamale, Ghana
- Karamandaneio Children's Hospital, Pátrai, Greece
- Tejasvini Hospital and Shantharam Shetty Institute of Orthopaedics and Traumatology (SSIOT) (Orthopaedics), Mangalore, India
- Lady Reading Hospital, Peshawar, Pakistan
- Spain (2):
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Universitario del Río Hortega, Valladolid
- Hospital Universitario de Caracas, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zomar BO, Chen M, Schaeffer EK, Mulpuri K, Joeris A; PedORTHO Study Group. Management of long bone fractures and traumatic hip dislocations in paediatric patients: study protocol for a prospective global multicentre observational cohort registry. BMJ Open. 2024 Mar 8;14(3):e079836. doi: 10.1136/bmjopen-2023-079836. PMID 38458811